CLINICAL TRIAL: NCT05189184
Title: Study of Camrelizumab in Combination With Apatinib Mesylate Plus Albumin-bound Paclitaxel and Cisplatin as the First Line Treatment of Recurrent or Metastatic, UnresectableHead and Neck Squamous Cell Carcinoma
Acronym: HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hong Zong, Chief physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSCC-R/M-01
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Inductive therapy with Camrelizumab and Apatinib Plus Albumin-bound paclitaxel and cisplatin
  Interventions: Drug: Camrelizumab+Apatinib mesylate+Albumin-bound paclitaxel+cisplatin

INTERVENTIONS:
Drug: Camrelizumab+Apatinib mesylate+Albumin-bound paclitaxel+cisplatin — Camrelizumab in Combination With Apatinib mesylate Plus Albumin-bound paclitaxel and cisplatin as the First Line Treatment of Recurrent or Metastatic , UnresectableHead and Neck Squamous Cell Carcinoma (HNSCC)

SUMMARY:
This is a prospective, open-labelled study to evaluate the efficacy and safety of Camrelizumab in Combination With Apatinib mesylate Plus Albumin-bound paclitaxel and cisplatin as the First Line Treatment of Metastatic or Recurrent, UnresectableHead and Neck Squamous Cell Carcinoma. The objective response rate (ORR) will be evaluated as the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1、Has fully understood and voluntarily signed an written Informed Consent and agreed to follow the research plan treatment and visiting plan; 2、Aged >=18 years; 3、Histologically confirmed recurrent or metastatic HNSCC of the oral cavity, oropharynx, hypopharynx, and/or larynx that is considered incurable by local therapies； 4、Eastern Cooperative Oncology Group (ECOG) performance status 0-1; 5、Expected survival period ≥ 3 months； 6、Tumor tissue with PD-L1 detection (paraffin specimens or fresh tumor tissue within 2 years) can be provided or PD-L1 test report of tumor tissue samples issued by a state-approved qualification unit； 7、At least one measurable lesion, according to RECIST 1.1; 8、Toxicity of the subject has been restored to the ≤1 level defined by NCI-CTCAE V5.0 (except hair loss)； 9、Patients must be able to swallow oral drugs and do not have significant affected gastrointestinal abnormalities, such as absorption adverse syndrome or most of the gastrointestinal tract; 10、The main function is normal, the test results at the time of screening must meet the following requirements:

1. Blood routine (no blood transfusion, erythropoietin (EPO), granulocyte-colony-stimulating factor (G-CSF) or granulocyte-macrophage-colony-stimulating factor (GM-CSF) within 14 days prior to screening) :

   A.Hemoglobin (HB) ≥ 90 g / L; B.Absolute neutrophil count (ANC) of >= 1.5*10^9/L； C.platelet count of >= 100*10^9/L；
2. Biochemical examination needs to meet the following criteria:

   A.TBIL < 1.5 ULN (Gilbert syndrome patient, < 3 ULN); B.ALT and AST < 3 ULN, if there exists hepatic metastases, ALT and AST < 5 ULN； C.Cr <=1.5 ULN or CCr ≥50ml/min;
3. Echocardiography：LVEF≥50%；
4. INR or PT <= 1.5 ULN, APTT <=1.5 ULN； 11、Contraception: Women of childbearing age should agree to use effective contraception during the study and for 6 months after the end of the study; Negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating; Men who agreed to use contraception during the study period and for six months after the end of the study period.

Exclusion Criteria:

1. Those who are allergic to drug treatment;
2. Disease that is suitable for local therapy administered with curative intent；
3. Accept system chemotherapy, but does not include a circulation of a multi-mode treatment for chemotherapy for local advanced diseases (this treatment end time must be 6 months from the first test for the first test);
4. Patients with local advanced head and neck squamous cell carcinoma have completed multi-mode chemotherapy completed within 6 months of disease progression;
5. It has received immunotherapy for anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody or targeted to T cell common stimulation or immunoction point pathway;
6. There have been any malignant tumors in five years, except for other malignant tumors,cervical in situ cancer, non-melanoma skin cancer or other tumors / cancer that passively treats for at least 5 years without disease;
7. Anti-blood vessel treatment was received within 6 months before administration;
8. According to NCI CTCAEV5.0, there have been peripheral neuropathy ≥ 2;
9. Accompanied by known active central nervous system transfer (CNS) and / or cancer meningitis: Previously received brain transfer subjects can participate in research, premise is the clinical stability for at least 2 weeks, no new or expanded brains Transfer evidence, and 14 days before the drug administration, steroids were stopped 14 days. The stable brain transfer in this definition should be determined before the study of drugs for the first time. The invisible brain transfer subject (ie there is no nervous system symptoms, no corticosteroids, no lesions> 1.5 cm) can participate, but need to periodically perform brain imaging in the disease site;
10. It has not been recovered from any acute impact of past surgery, chemotherapy or radiotherapy, ie, the subject of ≤1 (NCI CTCAEV5.0) (except for external hair loss), if the nutritional state is stable, it is allowed to radiotherapy and / or surgery Produced chronic advanced toxicity (pharyngeal / throat, namely oral dry, speech, swallowing abnormal)；
11. Within 4 weeks or 4 weeks before the first administration, the anti-tumor drug treatment (such as chemotherapy, hormone therapy, immunotherapy, antibody treatment, radiotherapy, etc.), except for reducing pain on bones, except for bones;
12. It has received major surgery within the 4 weeks of the first administration or is expected to carry out major surgery during this study;
13. In the first 2 weeks or 2 weeks of the first administration, immunosuppressive drugs is required, and the following is eliminated:

    1. intranasal, inhalation, external use steroids or local steroid injection (such as joint internal injection);
    2. physiological doses of systemic corticosteroids (≤10 mg / connone or equivalent dose);
    3. A short-term (≤7 days) use steroids to prevent or treat non-autoimmune allergic diseases; 14.、Subjects that are known to have active, or have a medical history and may relapse (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, Patients with multiple hardening, vascular, glomerulitis, etc.), or high risk (such as receiving organ transplantation require immunotherapy). However, the following patients are allowed to be incorporated: patients with type I diabetic patients with fixed doses; only the autoimmune thyroid dysfunction of hormone replacement treatment; skin disease (such as eczema, occupancy) without systemic treatment 10% or less ramp, no opaque symptoms of psoriasis, etc.); 15、15. There is a significant clinical cardiovascular disease, including but not limited to acute myocardial infarction within 6 months of the group, severe / unstable angina or coronary and bridge; congestive heart failure New York Heart Association (NYHA) ≥ 2 Level; arrhythmia (including QTC inter-male male ≥ 450 ms, female ≥ 470 ms); left ventricular ejection fraction (LVEF) <50%;

16、Under anti-hypertension treatment, still uncontrolled hypertension, defined as: systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg; 17、Urinalysis shows urine protein ≥2+ or 24-hour protein quantity test shows urinary protein ≥1 g; 18、History of mental drug abuse and unable to quit or have mental disabilities; 19、Active or uncontrolled severe infection; 20、It is known that there is a history of liver disease, including but not limited to known moonitis virus (HBV) infection and HBV DNA positive (≥1 × 104 copy / ml); Hepatitis Hepatitis Virus infection (HCV) and HCV RNA positive (≥1 × 103copy / ml), or cirrhosis, etc .; 21、Patients with pulmonary fibrosis, interstitial pneumonia, dust lung, radioactive pneumonia, drug-based pneumonia and severe lung function; 22、Pregnancy (pregnancy detection of pregnancy) or women underwater; 23、The first use of medication within 30 days or expected to vaccinate the vaccination during the study; 24、Subjects have or plans to receive physical organs or blood system transplants during the study (except corneal transplantation); 25、According to the judgment of the researcher, it is considered that it is not suitable for the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (CR+PR) | Time Frame: Up to 24 months
  Objective response rate (ORR) according to RECIST1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
Progression free survival (PFS) | Up to 24 months
  Progression free survival (PFS) according to RECIST 1.1

IPD SHARING:
Plan to Share IPD: No